CLINICAL TRIAL: NCT06164548
Title: Celiac Disease Among Egyptian Children With Unexplained Short Stature
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Esraa Atef Shehataa, 71515,Assiut, Assiut University
Other Study IDs: celiac disease
Record Dates: First submitted 2023-12-02; First posted 2023-12-11 (Actual); Last update posted 2023-12-11 (Actual); Status verified 2023-12

CONDITIONS: Celiac Disease
MeSH Terms: conditions — Celiac Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Detect the prevalence of celiac disease in children with unexplained short stature attended at Assiut University Children Hospital.

DETAILED DESCRIPTION:
Short stature is a term applied to a child whose height is 2 standard deviations or more below the mean for children of that chronological age and sex , and ideally of the same racial - ethnic group.This corresponds to a height below 3rd centile .Short stature can be the result of normal growth variants e.g. familial or constitutional which are the most common causes in children below one or two years ,or it can be the result of chronic systemic disorders, endocrine disorders, genetic, chromosomal disorders, and skeletal dysplasia. Chronic malnutrition and chemotherapy can also result in short stature -Around 3-2.5% of the children worldwide are short.

The Egyptian Demographic and Health Survey of 2008 (EDHS 2008) revealed that the prevalence of stunting among children under 5 was 2%28.9, while that of the EDHS 2014 was found to be 21%

* The goal of the evaluation of a child with short stature is to identify the subset of children with pathologic causes (such as Turner syndrome, inflammatory bowel disease , Celiac disease or other underlying systemic disease, or growth hormone deficiency). The evaluation also assesses the severity of the short stature and likely growth trajectory, to facilitate decisions about intervention, if appropriate.
* Celiac disease , also known as gluten enteropathy, is a chronic autoimmune condition, in genetically susceptible persons, perpetuated by the ingested gluten from cereals, wheat and barley,causes damage to the intestinal mucosa by an autoimmune reaction leading to villous atrophy. Villous atrophy then leads to multiple micro and macronutrient deficiencies.

Worldwide, its prevalence is about 1% ,affecting females twice more than males.

* Classic symptoms include gastrointestinal problems such as chronic diarrhea, abdominal distension, malabsorption, loss of appetite, and among children failure to grow normally. This often begins between six months and two years of age. Non-classic (extra intestinal) symptoms (eg, short stature, delayed puberty, epilepsy, peripheral neuritis and iron defiency anemia) are the most common, especially in people older than two years.
* Malabsorption is the typical presentation in early childhood, whereas older children with celiac disease can present with extra-intestinal symptoms including short stature and delay in pubertal development.

Short stature is the most commonly encountered extra- intestinal manifestation of CD in children, being found in roughly one-third of all new pediatric celiac diagnoses.

* Singh et al., showed an 11% prevalence of celiac disease among children presenting with short stature at a tertiary care hospital. Results from two European studies on short stature show celiac disease prevalence at 2:180 and 0:149 respectively. In short stature children without gastrointestinal signs, the prevalence of celiac disease raised up to 8-2%. By excluding endocrine causes of short stature, celiac disease prevalence will raise to even 59%
* In Egypt celiac disease is a frequent disorder among children, both in the general population (0.53%) and in at-risk groups (6.4%) The standard method of diagnosing celiac disease in symptomatic persons older than 2 years is the tissue transglutaminase (tTG) IgA test, followed by intestinal biopsy for histologic confirmation -The only known effective treatment is a strict lifelong gluten- free diet, which leads to recovery of the intestinal mucosa, improves symptoms, and reduced risk of developing complications in most people. If untreated it may result in cancers such as intestinal lymphoma and a slight increased risk of early death Vitamin and mineral supplements ,medications to control intestinal inflammation as steroids and Other drugs, such as azathioprine (Azasan, Imuran) or budesonide (Entocort EC, Uceris), might be used , in addition to control of complications like peripheral neuropathy, mouth ulcers and ataxia.

ELIGIBILITY:
Inclusion Criteria:

(1) Children aged between 2-18 years with undetectable causes of short stature whose height was < -2 SDfor the ageandsexaccording to Z score growth references for Egyptianchildrenand adolescent growth reference and Control DiseaseCenter(CDC) charts. (2) Short children not previously screened for Celiac disease.

Exclusion Criteria:

Short children with demonstrable cause such as:

(1) Familial and constitutional short stature. (2) Chronic illness. (3) Disproportionate short stature. (4) Short stature of endocrinal origin (eg, growth hormone deficiency). (5) Turner syndrome. (6) Short stature with significant congenital anomalies. (7) Patients on gluten free diet.

Ages: 2 Years to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: Children aged between 2-18 years with undetectable causes of short stature
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-01-15 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Celiac Disease Among Egyptian Children With Unexplained Short Stature | Baseline
  Detect prevalence of celiac disease in children presented with unexplained short stature

REFERENCES:
- [Background] Voss LD, Mulligan J, Betts PR, Wilkin TJ. Poor growth in school entrants as an index of organic disease: the Wessex growth study. BMJ. 1992 Dec 5;305(6866):1400-2. doi: 10.1136/bmj.305.6866.1400. PMID 1486305
- [Background] Ertekin V, Selimoglu MA, Kardas F, Aktas E. Prevalence of celiac disease in Turkish children. J Clin Gastroenterol. 2005 Sep;39(8):689-91. doi: 10.1097/01.mcg.0000174026.26838.56. PMID 16082278
- [Background] Ahmed ML, Allen AD, Sharma A, Macfarlane JA, Dunger DB. Evaluation of a district growth screening programme: the Oxford Growth Study. Arch Dis Child. 1993 Sep;69(3):361-5. doi: 10.1136/adc.69.3.361. PMID 7692826
- [Background] Itzlinger A, Branchi F, Elli L, Schumann M. Gluten-Free Diet in Celiac Disease-Forever and for All? Nutrients. 2018 Nov 18;10(11):1796. doi: 10.3390/nu10111796. PMID 30453686
- [Background] Jericho H, Sansotta N, Guandalini S. Extraintestinal Manifestations of Celiac Disease: Effectiveness of the Gluten-Free Diet. J Pediatr Gastroenterol Nutr. 2017 Jul;65(1):75-79. doi: 10.1097/MPG.0000000000001420. PMID 28644353